CLINICAL TRIAL: NCT00871052
Title: Calcipotriol in the Prevention of Polymorphic Light Eruption
Brief Title: Calcipotriol and Polymorphic Light Eruption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Peter Wolf, MD, Principal Investigator, Medical University of Graz, Austria
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Graz IRB 19-129 ex 07/08
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Polymorphic Light Eruption
Keywords: Polymorphic light eruption; UV radiation; Vitamin D; Immune suppression; Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Calcipotriol-containing cream — Topical treatment twice a day for 7 days
  Other Names: Vitamin D3 analogue

SUMMARY:
Polymorphic light eruption (PLE) is a photodermatosis with an extremely high prevalence, particularly among young women (up to 20%). The disease is characterized through itchy skin lesions on sun-exposed body sites occurring after sun exposure mostly in spring and early summer. Its etiopathogenesis is unknown but resistance to ultraviolet radiation (UVR)-induced immunosuppression with subsequent immune reactions against skin photoneoantigens has been suggested.

The phenomenon of UVR-induced immunosuppression (suppression of CHS) has been well known for many years. Recent findings showed that regulatory T cells (CD4+CD25+FoxP3+) (Tregs), a subset of T helper cells, are crucial in UVR-induced immunosuppression. However, the requirements for the maintenance of peripheral CD4+CD25+ T cells, important in suppression of immune responses, are still incompletely understood. Recent work suggests that cutaneous RANKL might be the physiologic missing link that couples UVR to immunosuppression. Epidermal RANKL, expressed in keratinocytes of inflamed skin due to e.g. UVR exposure was shown to control the number of Tregs via activation of dendritic cells, hereby mediating UVR-induced immunosuppression (e.g. suppression of allergic contact hypersensitivity responses). In addition to the suppression of local cutaneous hyperallergic responses, the development of systemic autoimmunity is suppressed. A strong inducer of RANKL expression and of Tregs is vitamin D3 that has been reported to have immunosuppressive effects. Interestingly, patients with autoimmune disorders (e.g. lupus erythematosus) may exhibit reduced vitamin D3 blood levels.

This randomized, double blinded left-right body side experimental comparison study was designed to assess the preventive effect of the vitamin D3 analogue calcipotriol in patients with PLE. The hypothesis is tested that treatment with a calcipotriol-containing cream can prevent the UVR-induced development of PLE skin lesions. Better insight into the pathogenesis of PLE may give clues to develop new therapeutic strategies.

DETAILED DESCRIPTION:
PLE patients will be recruited through the Photodermatology Unit of the Department of Dermatology, Medical University of Graz, Austria. Eligible patients will be identified through diagnosis-related computer-assisted search in the electronic patient chart system of the Unit. The diagnosis of PLE will be verified by patient's history, clinical symptoms, histologic findings, laboratory studies and/or phototesting procedures.

A calcipotriol-cream and a placebo cream are used in this study. Fifteen PLE patients will be enrolled. On day 1, the individual minimal erythema dose (MED) is assessed on patients' skin by exposure to a test ladder of solar-simulated UVR produced by a xenon arc source (Oriel Corp. Darmstadt, Germany). From day 2 to 5, 0.5 individual MED exposures (increased by 0 to 30% per exposure, depending on the erythema response to a preceding dose) are given to a total of four 10-by-10 cm skin test fields on symmetrically located, individual PLE predilection sites on the trunk or extremities. These test fields are pretreated in a randomized and double-blinded fashion either with the calcipotriol cream or the placebo cream (twice a day) during 7 days before start of phototesting.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PLE either by typical history and/or typical histology of lesions and/or positive phototesting results
* Age > 18 years

Exclusion Criteria:

* Presence of or history of malignant skin tumors
* Dysplastic melanocytic nevus syndrome
* Photosensitive diseases such as porphyria, chronic actinic dermatitis, Xeroderma pigmentosum, basal cell nevus syndrome, and others
* Autoimmune disorders such as Lupus erythematosus or dermatomyositis
* Psychiatric disorders
* Immune deficiency or systemic treatment with steroids and/or other immunosuppressive drugs
* Pregnancy or lactation
* Antinuclear antibodies
* UV exposure in test fields within 8 weeks before study start
* General poor health status
* Severe liver or renal disease, disorders or therapy of the calcium metabolism with vitamin D containing drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Polymorphic light eruption score | 2 weeks

SECONDARY OUTCOMES:
Pruritus | 2 weeks
Erythema | 2 weeks
Tanning | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wolf, MD, Principal Investigator — Medical University of Graz, Austria
Locations (1):
- Medical University, Department of Dermatology, Graz, Austria

REFERENCES:
- [Derived] Gruber-Wackernagel A, Bambach I, Legat FJ, Hofer A, Byrne SN, Quehenberger F, Wolf P. Randomized double-blinded placebo-controlled intra-individual trial on topical treatment with a 1,25-dihydroxyvitamin D(3) analogue in polymorphic light eruption. Br J Dermatol. 2011 Jul;165(1):152-63. doi: 10.1111/j.1365-2133.2011.10333.x. Epub 2011 May 30. PMID 21428979